CLINICAL TRIAL: NCT01623089
Title: Identification of Asthma Phenotypes in Severe Asthmatics
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2010/810/C
Record Dates: First submitted 2012-06-15; First posted 2012-06-19 (Estimated); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Asthma
Keywords: severe asthma, phenotype, data
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- severe asthma

SUMMARY:
Asthma is a heterogenous disease. Different patients have different presentations, course of disease and response to treatment.

The investigators would like to study our population of more severe asthma and find out about their profile - demographic, clinical and inflammatory.

DETAILED DESCRIPTION:
Asthma is a heterogeneous disorder presenting with many phenotypes. Most asthmatics have mild to moderate disease. However, 5-20% of asthmatics belong to the "Difficult-to-treat" or more severe group and they account for 50-80% of asthma health care costs. In a tertiary hospital like Singapore General Hospital, most of our asthmatics belong to the more severe group. They have more frequent healthcare visits, hospitalizations, medication use and higher risks of death.

There is currently no local data on the phenotypic profile of our patients. Asthma phenotypes which have been identified include those related to triggers ( eg. drugs such as aspirin or NSAIDS, environmental allergen, occupational allergens or irritants, exercise) or clinical physiological phenotypes ( eg. severity-defined, exacerbation-prone, chronic airflow limitation, steroid-resistant, age -of -onset) or inflammatory phenotypes ( eg. eosinophilic, neutrophilic, pauci granulocytic, mixed). With better understanding of their phenotypes, treatment can then be individually tailored to improve their asthma control and reduce future risks.

We aim to improve the understanding of this group of asthmatics such that better treatment approaches can be developed in the future. This is not a clinical trial. Its purpose is to gather information ranging from demographic data, medical history to responses to simple routine questions, to lung function, inflammation, allergy and blood testing results. The data are analyzed to improve our understanding of the clinical and inflammatory phenotypes ( or profiles) in this group of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Difficult-to-treat severe asthma
2. Treatment-resistant severe asthma patients who are partially or poorly controlled despite high dose inhaled corticosteroids ( ICS) or a high-dose ICS and long acting- beta-2- agonist combination ( LABA) and frequent or chronic use of systemic corticosteroids or
3. Treatment-resistant severe asthma who are well-controlled on the highest level of recommended treatment to maintain control (high dose ICS or combination of high-dose ICS with other medications such as LABA, theophylline, montelukast, systemic corticosteroids, anti-Ig E, etc.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Respiratory or severe asthma clinic
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2011-01-02 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Annual exacerbation rates | Through study completion, an average of 1 year
  Annual exacerbation rates
Symptom control | Through study completion, an average of 1 year
  Symptom control using Asthma Control Test

CONTACTS AND LOCATIONS:
Overall Officials: Mariko Koh, MBBS, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No